CLINICAL TRIAL: NCT05516381
Title: Evaluation of Navigation-Assisted TKA Using Mechanical vs. Restricted Kinematic Alignment on Patient Reported Outcome Measures (PROMs): A Prospective, Randomized Clinical Study
Brief Title: Evaluation of Navigation-Assisted TKA Using Mechanical vs. Restricted Kinematic Alignment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: TM-2021-1586
Record Dates: First submitted 2022-08-19; First posted 2022-08-25 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Knee Arthroplasty, Total

STUDY DESIGN:
Intervention Model Description: Randomization list (block randomized, computer generated, two equal-size groups) will be created within the EDC system
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study and research staff will be blinded to randomization and the cohort allocation until after consenting and eligibility is determined. Subjects will be blinded to the randomization (MA TKA or restricted iKA TKA) until the completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Restricted Invers Kinematic Knee Alignment Technique (Other): Restricted Invers Kinematic Knee Alignment Technique
  Interventions: Device: Optetrak Logic CR Knee System
- Mechanical Knee Alignment Technique (Other): Mechanical Knee Alignment Technique
  Interventions: Device: Optetrak Logic CR Knee System

INTERVENTIONS:
Device: Optetrak Logic CR Knee System — The OPTETRAK® Comprehensive Knee System consists of the OPTETRAK® Total Knee System and the OPTETRAK Logic® Total Knee System. The OPTETRAK Comprehensive Knee System comprises both non-porous and porous knee prostheses for use in total-knee joint replacement procedures. (In the USA, the OPTETRAK Comprehensive Knee System is indicated for cemented use only, except for the OPTETRAK Logic PS and CR Porous Femoral Components, which are indicated for cemented or cementless use.) The system includes various sizes and types of modular femoral components, tibial components, patellar components, and accessories for use in primary and revision applications.
  Other Names: Exactech Guided Personalized Surgery

SUMMARY:
The purpose of this study is to evaluate both clinical measures and PROMs in patients undergoing total knee arthroplasty (TKA) using restricted inverse kinematic alignment (iKA) compared to mechanical alignment (MA), both using surgical navigation assistance.

DETAILED DESCRIPTION:
A prospective randomized clinical study will be conducted.

The study will consist of two cohorts and will collect clinical data from a maximum of 148 knee arthroplasty surgeries during which the patient will receive the Optetrak Logic® CR TKA device. Cohorts will consist of 1) subjects undergoing MA TKA and 2) subjects undergoing restricted iKA TKA. All cohorts will utilize navigation-assisted surgery (ExactechGPS®) and will be enrolled and consented concurrently. Subjects will be randomized and have a 50% chance of being assigned to the MA TKA cohort and a 50% chance of being assigned to the restricted iKA TKA cohort. Study and research staff will be blinded to randomization and the cohort allocation until after consenting and eligibility is determined. Subjects will be blinded to the randomization (MA TKA or restricted iKA TKA) until the completion of the study.

Data collection under this protocol shall be conducted in a way that conforms to any applicable local and national rules, regulations, and guidelines relating to the conduct of clinical research and the protection of human subjects. As appropriate, this may include but is not limited to the following: Good Clinical Practice (GCP) requirements, FDA regulations and guidelines, ISO 14155: 2020, ICH guidelines, HIPAA and other regulations pertaining to the protection of patient data and data privacy, guidelines established by local Institutional Review Boards or similar Ethics Committees, the Belmont Report, and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be included in the study:

  1. Subject must be at least 18 years of age at the time of the surgery (skeletally mature)
  2. Subject will receive a Optetrak Logic® CR device per the "Indications for Use" described above
  3. Subject must be willing to comply with the pre-operative and post-operative visit requirements
  4. Subject must be willing and able to provide written informed consent for participation in the study

Exclusion Criteria:

* Subjects will be excluded from the study if they meet any of the following exclusion criteria:

  1. Subject with a suspected or confirmed systemic infection and/or a secondary remote infection
  2. Subject without sufficient bone stock to allow appropriate insertion and fixation of the prosthesis
  3. Subject without sufficient soft tissue integrity to provide adequate stability
  4. Subject with either mental or neuromuscular disorders that do not allow control of the knee joint
  5. Subjects whose weight, age, or activity level might cause extreme loads and early failure of the system
  6. Subject is participating in another drug or device study other than knee replacement within the last three (3) months
  7. Subject has behavioral and/or mental issues that may interfere with their ability to follow post-operative instructions
  8. Subject is a prisoner
  9. Subject is pregnant
  10. Subject is undergoing radiation therapy where the targeted field involves the knee joint
  11. Subjects with malignancy involving proximal tibia, distal femur, or knee joint
  12. Subjects undergoing active administration of chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score (KSS) | 3-month
  Validated outcome score
Knee Society Score (KSS) | 6-month
  Validated outcome score
Knee Society Score (KSS) | 12-month
  Validated outcome score
Forgotten Joint Score (FJS) | 3-month
  Validated outcome score
Forgotten Joint Score (FJS) | 6-month
  Validated outcome score
Forgotten Joint Score (FJS) | 12-month
  Validated outcome score
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 3-month
  Validated outcome score
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 6-month
  Validated outcome score
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 12-month
  Validated outcome score
Visual Analog Scale (VAS) - Pain | 3-month
  Visual scale from 1-10 (low score is better)
Visual Analog Scale (VAS) - Pain | 6-month
  Visual scale from 1-10 (low score is better)
Visual Analog Scale (VAS) - Pain | 12-month
  Visual scale from 1-10 (low score is better)
Visual Analog Scale (VAS) - Patient Satisfaction | 3-month
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Patient Satisfaction | 6-month
  Visual scale from 1-10 (high score is better)
Visual Analog Scale (VAS) - Patient Satisfaction | 12-month
  Visual scale from 1-10 (high score is better)

SECONDARY OUTCOMES:
Knee Alignment | Intraoperative
  Characterization of knee in terms of ligament balancing will be assessed through constant-pressure full arc of motion measurement.

CONTACTS AND LOCATIONS:
Overall Officials: David Mateu-Vincent, Medical Degree, Principal Investigator — Orthpaedic Surgeon Hospital Universitaria Mutua Terrassa
Locations (1):
- Fundacio Mutua de Terrassa per a la Docenia i Recera Biomedica i Social, F.P.C., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data

REFERENCES:
- [Background] Winnock de Grave P, Luyckx T, Claeys K, Tampere T, Kellens J, Muller J, Gunst P. Higher satisfaction after total knee arthroplasty using restricted inverse kinematic alignment compared to adjusted mechanical alignment. Knee Surg Sports Traumatol Arthrosc. 2022 Feb;30(2):488-499. doi: 10.1007/s00167-020-06165-4. Epub 2020 Jul 31. PMID 32737528
- [Background] Almaawi AM, Hutt JRB, Masse V, Lavigne M, Vendittoli PA. The Impact of Mechanical and Restricted Kinematic Alignment on Knee Anatomy in Total Knee Arthroplasty. J Arthroplasty. 2017 Jul;32(7):2133-2140. doi: 10.1016/j.arth.2017.02.028. Epub 2017 Feb 20. PMID 28302462